CLINICAL TRIAL: NCT03453424
Title: Analgesic Efficacy of Dexmedetomidine Added to Patient Controlled Epidural Analgesia for Patients Undergoing Major Abdominal Cancer Surgery
Brief Title: Analgesic Efficacy of Dexmedetomidine Added to Fentanyl in PCEA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Alaa Ali M. Elzohry, Principal Investigator, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SECI
Record Dates: First submitted 2018-02-21; First posted 2018-03-05 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Abdominal Pain; Abdominal Cancer
MeSH Terms: conditions — Abdominal Pain | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEA+DEX group (Active Comparator): Intra operative thoracic epidural injection of (bupivacaine 0.125% +fentanyl 2 mic/ ml) , initial bolus dose of 8 ml before skin incision followed by fixed rate infusion of 6 ml/h till end of abdominal layer closure.
  Postoperative, thoracic epidural injection of (bupivacaine 0.0625%+fentanyl 2 mic /ml + dexmedetomidine 0.5 mic/ ml) at infusion rate 6 ml /h and bolus dose of 3 ml with lockout time 10 min
  Interventions: Procedure: TEA+DEX
- TEA group (Active Comparator): Intraoperative,thoracic epidural injection of bupivacaine (0.125%+fentanyl 5 mic/ml ) ,initial bolus dose of 8 ml before skin incision followed by fixed rate infusion of 6 ml/h till start of abdominal layer closure.
  Postoperative, thoracic epidural injection of (bupivacaine 0.0625%+fentanyl 2 mic /ml) at infusion rate 6 ml /h and bolus dose of 3 ml with lockout time 10 min
  Interventions: Procedure: TEA

INTERVENTIONS:
Procedure: TEA+DEX — intra and post operative TEA infusion of (bupivacaine +fentanyl 2 mic/ ml+ dexmedetomidine 0.5 mic/ ml) Under strict aseptic precautions thoracic epidural was performed using a 16 gauge,Tuhy epidural needle by a paramedian approach. T8-T9 inter space was chosen for the injection. Skin at insertion site was anesthetized by 3 ml of lidocaine 1%, the epidural space was identified by the loss of resistance technique, the catheter was introduced approximately 2-4 cm into the epidural space, epidural test dose consisted of 3 ml of lidocaine 2 % with 1: 200,000 adrenaline.
  Arms: TEA+DEX group
Procedure: TEA — Under strict aseptic precautions thoracic epidural was performed using a 16 gauge,Tuhy epidural needle by a paramedian approach. T8-T9 interspace was chosen for the injection. Skin at insertion site was anesthetized by 3 ml of lidocaine 1%, the epidural space was identified by the loss of resistance technique, the catheter was introduced approximately 2-4 cm into the epidural space, epidural test dose consisted of 3 ml of lidocaine 2 % with 1: 200,000 adrenaline.
  then, intra and post operative TEA infusion of bupivacaine 0.125%+fentanyl 2 mic/ ml.
  Arms: TEA group

SUMMARY:
Dexmedetomidine if add to patient controlled epidural analgesia for patients undergoing major abdominal cancer surgery may improve its effects.

DETAILED DESCRIPTION:
The aim of modern anaesthetic practice is to insure the rapid recovery of patients with fewer complications and earlier hospital discharge.

Thoracic epidural anesthesia (TEA) has been established as a cornerstone in the perioperative care after thoracic and major abdominal surgery providing most effective analgesia. beyond its analgesic properties, TEA's effects on the postoperative neurohumoural stress response, cardiovascular Pathophysiology, and intestinal dysfunction have been in the focus of both clinical and experimental investigations for years.

dexmedetomidine if add to patient controlled epidural analgesia for patients undergoing major abdominal cancer surgery may improve its effects.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (21 years old or more),
* classified as American Society of Anesthesiologists (ASA) grade II and III,
* scheduled for elective major abdominal cancer surgery.

Exclusion Criteria:

* patients with coagulopathy,
* active neurological disease,
* cutaneous disorders at the epidural insertion site,
* allergy to the study medication
* and patients refusal.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change in pain scores (dynamic VAS) | at 0, 4, 8, 12, 18, 24, 36 and 48 hours post operative.
  dynamic visual analogue scale (0-10) 0=no pain 10=worst imaginable pain

SECONDARY OUTCOMES:
Change in post operative MAP | at 0, 4, 8, 12, 18, 24, 36 and 48 hours post operative.
  Mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M. Elzohry, MD, Principal Investigator — Lecturer in Assuit university
Locations (1):
- South Egypt Cancer Institute, Assiut University, Arab Republic of Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No